CLINICAL TRIAL: NCT00037986
Title: Functioning, Disability, and Quality of Life in the Adult Hearing Impaired
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Abrams, Harvey - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2439R
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Hearing Impaired
Keywords: Audiology; Hearing; Hearing Aids; Quality of Life
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

ARMS (1):
- 1 (Other)
  Interventions: Device: Hearing Aids

INTERVENTIONS:
Device: Hearing Aids — Hearing aid use

SUMMARY:
The short-term research objectives of the proposed study are as follows:

1. To measure the effects of audiological intervention on selected domain specific (i.e., Communicative, Interpersonal, and Social roles) and overall functioning using the WHO-DASII, a generic health measure conceptually grounded in the ICIDH-2 model of disablement and functioning.
2. To measure the effects of audiological intervention on selected domain specific (i.e., Role Functioning-Emotional; and, Social Functioning) and overall functioning using the MOS-SF36V, a generic health measure currently utilized in the Veteran's Health Administration.
3. To determine the accuracy with which measures of audibility (SII), hearing handicap (HHIE), and, hearing disability (APHAB) predict domain specific and overall functioning, and life-satisfaction as measured by the WHO-DASII and the MOS-SF36V will be evaluated.
4. To compare hearing aid treatment effects as measured by changes in WHO-DASII domain specific and overall functioning scores to those measured by changes in disease specific instruments examining similar constructs.
5. To compare hearing aid treatment effects as measured by changes in MOS-SF36V domain specific and overall functioning scores to those measured by changes in disease specific instruments examining similar constructs.
6. To determine and compare cost-effectiveness of hearing aid intervention as calculated using WHO-DASII and MOS SF-36V outcome data.

The long-term research objective is to compare the cost-effectiveness and cost-utility of audiologic intervention with those of other health care interventions commonly associated with the veteran population (e.g. mental health, cardiology, pulmonary, orthopedic, etc.).

DETAILED DESCRIPTION:
Specific Objectives with Projected Timetable:

1. . Short-term objectives:

   1. . To measure the effects of audiological intervention on selected domain specific (i.e., Communicative, Interpersonal, and Social roles) and overall functioning using the WHO-DAS II, a generic health measure conceptually grounded in the International Classification of Impairment, Disability, and Handicap (ICIDH)-2 model of disablement and functioning (WHO, 1999).
   2. . To measure the effects of audiological intervention on selected category specific (i.e., Role Functioning-Emotional and Social Functioning) and overall functioning using the MOS-SF36V, a generic health measure currently utilized in the Veterans Health Administration.
   3. . To determine the accuracy with which measures of audibility (SII), hearing handicap (HHIE), and, hearing disability (APHAB) predict domain specific and overall functioning, and life-satisfaction as measured by the WHO-DAS II and the MOS-SF36V will be evaluated.
   4. . To compare hearing aid treatment effects as measured by changes in WHO-DAS II domain specific and overall functioning scores to those measured by changes in disease specific instruments examining similar constructs.
   5. . To compare hearing aid treatment effects as measured by changes in MOS-SF36V domain specific and overall functioning scores to those measured by changes in disease specific instruments examining similar constructs.
   6. . To determine and compare cost-effectiveness of hearing aid intervention as calculated using WHO-DAS II and MOS-SF36V outcome data.
2. . Long-term objective: To compare the cost-effectiveness and cost-utility of audiologic intervention with those of other health care interventions commonly associated with the veteran population (e.g. mental health, cardiology, pulmonary, orthopedic, etc.).

ELIGIBILITY:
Inclusion Criteria:

Hearing impaired

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2001-07; Primary Completion 2004-05 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
WHO-DAS II | 2, 6, and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Abrams, PhD, Principal Investigator — VA Medical Center, Bay Pines
Locations (1):
- VA Medical Center, Bay Pines, Bay Pines, Florida, United States

REFERENCES:
- [Result] Abrams HB, Chisolm TH, McArdle R. Health-related quality of life and hearing aids: a tutorial. Trends Amplif. 2005;9(3):99-109. doi: 10.1177/108471380500900302. PMID 16244757
- [Result] McArdle R, Chisolm TH, Abrams HB, Wilson RH, Doyle PJ. The WHO-DAS II: measuring outcomes of hearing aid intervention for adults. Trends Amplif. 2005;9(3):127-43. doi: 10.1177/108471380500900304. PMID 16244759
- [Result] Chisolm TH, Abrams HB, McArdle R, Wilson RH, Doyle PJ. The WHO-DAS II: psychometric properties in the measurement of functional health status in adults with acquired hearing loss. Trends Amplif. 2005;9(3):111-26. doi: 10.1177/108471380500900303. PMID 16244758